CLINICAL TRIAL: NCT04735614
Title: The Effect of Physical Thoracic Stabilization on Pain Control in Patients Who Had a Lung Tumor and Received Video-assisted Thoracoscopic Surgery: A Randomized Controlled Trial.
Brief Title: Physical Stabilization in Post-VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 109-118-F
Record Dates: First submitted 2021-01-19; First posted 2021-02-03 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer; Pain, Postoperative
Keywords: video-assisted thoracoscopic surgery; VATS; post-operation pain control; patient-controlled analgesia; visual analogue scale; Posthorax Thoraxbelt
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon will not know the patients' group before or during the surgery. The outcome assessor won't know the group during the whole research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ThoraxBelt (Experimental): Received ThoraxBelt after the surgery. Standard care for pain management will be the same as the Standard Care Arm.
  Interventions: Device: Posthorax Thoraxbelt
- Standard care (No Intervention): Standard care with IV PCA and on-request oral painkiller.

INTERVENTIONS:
Device: Posthorax Thoraxbelt — The patients will be assisted to put on the ThoraxBelt after the surgery by our research member and will be asked to keep it on except for during showering through the whole study period.
  Arms: ThoraxBelt

SUMMARY:
Background: Post-video-assisted thoracic surgery (VATS) pain remains an open issue, though most patients experience less acute pain after VATS than thoracotomy. So far, there was no gold standard regarding pain control post-VATS.

Objective: To conduct a randomized controlled trial assessing the effect of physical thoracic stabilization on post-VATS pain control.

Method: The investigators aimed to recruit 40 patients with operable lung cancer in the outpatient clinic from January to December 2021. The patients will be randomized into the intervention or control group. The intervention group will receive physical thoracic stabilization with POSTHORAX ThoraxBelt after the surgery, whereas the control group will have standard care. The follow-up period will last for 6 months.

DETAILED DESCRIPTION:
The study has been approved by the hospital research ethics committee.

Arm 1: Physical thoracic stabilization with ThoraxBelt after VATS Arm 2: Standard care after VATS

Primary outcome: Visual analog scale (VAS) 6 hours, 24 hours, and 48 hours after the surgery.

Secondary outcomes:

1. The accumulated dose of the intervenous patient-controlled analgesic drug.
2. The dose of oral painkiller administered during the hospital stay.
3. Complications related to the ThoraxBelt.
4. Hospital stay
5. VAS before discharge
6. Unanticipated events (ICU admission, a second surgery, death)
7. VAS during the 2-week, 1-month, 2-month, 6-month outpatient clinic visit after the surgery.
8. Compliance on ThoraxBelt.

ELIGIBILITY:
Inclusion Criteria:

* Operable lung cancer
* Eligible for video-assisted thoracoscopic surgery

Exclusion Criteria:

* Known allergy to ThoraxBelt
* Chest wall Infection or other diseases
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale(VAS) | 48 hours
  A pain score will be assigned to each patient after the total amount of visual analog scale. The minimum is 0 and the maximum is 10, which 10 indicated the most pain.

SECONDARY OUTCOMES:
IV PCA dose | 48 hours
  the accumulated IV PCA drug dose
On-request oral painkiller dose | 48 hours
  the accumulated oral painkiller dose
Complications during hospital stay | 48 hours
  Any complications related to ThoraxBelt or not
Length of hospital stay | 1 month
  The number of days in the hospital stay.
The number of unanticipated events | 1 month
  The number of unanticipated events including ICU admission, a second surgery or death will be documented in both groups.
Visual analog scale in outpatient clinic follow-up | 6 months
  follow-up 2-week, 1-month, and 6-month after discharge. The minimum is 0 and the maximum is 10, which 10 indicated the most pain.
Compliance of ThoraxBelt after discharge | 2 months
  How long is the ThoraxBelt removed except during bath in a day. The unit is hour.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently, we have no plan on sharing the IPD.

REFERENCES:
- [Derived] Fan CY, Lin CW, Sung CW, Huang EP. Therapeutic potential of physical stabilization in VATS pain control: a randomized controlled trial. Updates Surg. 2025 Jan;77(1):193-199. doi: 10.1007/s13304-024-01999-w. Epub 2024 Sep 15. PMID 39277837